CLINICAL TRIAL: NCT03870893
Title: Effects of Hippotherapy on Physical Activities, Cardiopulmonary Fitness and Attention in Children With Cerebral Palsy
Brief Title: Effects of Hippotherapy on Physical Fitness and Attention in Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Collaborators: National Research Foundation of Korea (Other)
Responsible Party: Principal Investigator, Jeong Yi Kwon, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2017-0665-000
Record Dates: First submitted 2017-07-26; First posted 2019-03-12 (Actual); Results first posted 2020-08-05 (Actual); Last update posted 2020-08-05 (Actual); Status verified 2020-07

CONDITIONS: Cerebral Palsy; Physical Activity; Attention Disorder
Keywords: cerebral palsy; hippotherapy; cardiopulmonary fitness; physical activity; attention
MeSH Terms: conditions — Cerebral Palsy; Motor Activity; Cognition Disorders | interventions — Equine-Assisted Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention is administered to patients in this Arm.
  Interventions: Behavioral: hippotherapy
- control group (No Intervention): No intervention

INTERVENTIONS:
Behavioral: hippotherapy — 16weeks hippotherapy program
  Arms: Intervention group

SUMMARY:
This research analyzes whether hippotherapy improves the physical activity, cardiopulmonary fitness, and attention in children with cerebral palsy and whether this enhances their general health and quality of life.

DETAILED DESCRIPTION:
This research aims to promote hippotherapy by scientifically proving its therapeutic effects and mechanism to contribute to improving the health and quality of life of the patients as well as reducing their global burden of disease by shifting the current passive "therapy-oriented" paradigm to a more proactive "participation-oriented" paradigm.

Ever since physical activity and physical fitness have been reported to have an inverse relationship with the mortality rate, especially deaths due to cardiovascular disease, various efforts have been made to optimize physical activity and physical fitness among children with cerebral palsy. ADHD is one of the most common coexisting conditions of cerebral palsy. More participation in engaging sports activities like therapeutic riding is anticipated to improve patient health and their quality of life.

Hippotherapy is expected to improve clinical symptom of ADHD in children with cerebral palsy while preventing possible ensuing psychiatric disorders, thereby bringing significant improvement in their health and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of spastic CP
* GMFCS level I-III
* weight < 35kg
* ability to walk independently with or without an assistive device
* ability to comply with the study protocol and follow verbal directions

Exclusion Criteria:

* botulinum toxin injection within 3 months
* orthopedic surgery within 1 year (difficulty performing one step instructions)
* moderate to severe intellectual disability
* uncontrolled seizure
* poor visual or hearing acuity
* patients who weigh more than 35 kg
* hip dislocation
* scoliosis more than 30 degrees
* musculoskeletal surgery within 1 year

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 47 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minhwa Suk, Principal Investigator — Researcher
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Suk MH, Kwon JY. Effect of Equine-Assisted Activities and Therapies on Cardiorespiratory Fitness in Children with Cerebral Palsy: A Randomized Controlled Trial. J Integr Complement Med. 2022 Jan;28(1):51-59. doi: 10.1089/jicm.2021.0158. PMID 35085017
- [Derived] Ahn B, Joung YS, Kwon JY, Lee DI, Oh S, Kim BU, Cha JY, Kim JH, Lee JY, Shin HY, Seo YS. Effects of equine-assisted activities on attention and quality of life in children with cerebral palsy in a randomized trial: examining the comorbidity with attention-deficit/hyperactivity disorder. BMC Pediatr. 2021 Mar 19;21(1):135. doi: 10.1186/s12887-021-02597-0. PMID 33740922
- [Derived] Park IK, Lee JY, Suk MH, Yoo S, Seo YG, Oh JK, Kwon JY. Effect of Equine-Assisted Activities on Cardiac Autonomic Function in Children with Cerebral Palsy: A Pilot Randomized-Controlled Trial. J Altern Complement Med. 2021 Jan;27(1):96-102. doi: 10.1089/acm.2020.0346. Epub 2020 Nov 27. PMID 33252241

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention Group: Children participated in Hippotherapy for 40 minutes per lesson twice a week for 16 weeks (total of 32 sessions).
Period: Overall Study
Arm/Group | Intervention Group | Control Group
Started | 23 | 24
Completed | 23 | 23
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention Group | Control Group | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 23 | 23 | 46
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.74 (1.63) | 7.22 (1.48) | 7.48 (1.56)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 12 | 12 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 23 | 23 | 46
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  South Korea | 23 | 23 | 46

OUTCOME MEASURES:

1. Primary Outcome: Change of Clinical Global Improvement(CGI)
Description: The Clinical Global Impression - Severity scale (CGI-S) is a 7-point scale that requires the clinician to rate the severity of the patient's illness at the time of assessment, relative to the clinician's past experience with patients who have the same diagnosis. Possible ratings are 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients. Lower values represent a better outcome.
  The Clinical Global Impression - Improvement scale (CGI-I) is a 7 point scale that requires the clinician to assess how much the patient's illness has improved or worsened relative to a baseline state at the beginning of the intervention. and rated as 1= very much improved; 2=much improved; 3=minimally improved; 4=no change; 5=minimally worse; 6=much worse; 7=very much worse. Higher values represent a better outcome.
Time Frame: Change in baseline CGI at 16weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
score on a scale
  Change of CGI-S | -0.13 (0.46) | -0.09 (0.29)
  Change of CGI-I | 2.65 (0.78) | 3.87 (0.46)

2. Secondary Outcome: Change of Attention
Description: Child Behavior Checklist; The Social Ability Scale consists of Sociality Scale and Academic Performance Scale. The Scale of Problem Behavior Syndrome consists of 113 items related to problem behavior, and 13 (Sociality, Learning Problem, Total Social Ability, Atrophy, Depression, social immaturity, thinking problems, attention problems, flying, aggression, internalization problems, externalizing problems, total problem behaviors). For each question, the scale is to be rated as 3-point Likert scale, the raw scores of all subscales are converted to standardized T scores . The higher the score, the higher the tendency toward problem behavior.
Time Frame: Change in baseline attention at 16weeks
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
T-score
  Total problems(pre) | 57.52 (9.08) | 57.70 (7.15)
  Total problems(post) | 54.61 (11.63) | 55.39 (7.55)

3. Secondary Outcome: Change of Physical Activity(%)
Description: The %sedentary physical activity(%SPA), %light physical activity(%LPA), %moderate physical activity(%MPA), %vigorous physical activity(%VPA) during the day using ActiGraph(model GT3X, ActiGraph, Pensacola, FL, USA).
Time Frame: Change in baseline physical activity at 16weeks
Measure: Mean (Standard Deviation); unit: percentage of physcal activity
Groups:
- Intervention Group: Children participated in Hippotherapy for 40 minutes per lesson twice a week for 16 weeks (total of 32 sessions) in addition to conventional physiotherapy.
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
percentage of physcal activity
  Change of %SPA | 1.86 (5.07) | -0.61 (4.86)
  Change of %LPA | -1.58 (4.41) | 0.24 (3.74)
  Change of %MPA | -0.28 (0.67) | 0.13 (1.00)
  Change of %VPA | 0.00 (0.53) | 0.25 (0.75)

4. Secondary Outcome: Change of Peak Oxygen Uptake(VO2peak)
Description: peak oxygen uptake(ml/kg/min) is a category of physical fitness, which is measured during graded submaximal exercise test. Higher values represent a better outcome.
Time Frame: Change in baseline peak oxygen uptake at 16weeks
Population: Five Participants want to stop during measurement (Intervention group -> 3 participants; Control group -> 2 participants)
Measure: Mean (Standard Deviation); unit: ml/kg/min
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 21
ml/kg/min | 1.84 (4.33) | -0.09 (3.57)

5. Secondary Outcome: Change of Gross Motor Function Measure 66
Description: GMFM-88 is a measure developed to evaluate the gross motor function changes in CP children. It has five components: lying and rolling, sitting, kneeling and crawling, standing, and walking. The score of each dimension is expressed as a percentage of the maximum score. The GMFM-66, which includes 66 items of the original 88 items. Item scoring is the same for the GMFM-88 and the GMFM-66. There is a scoring system with each item scored as 0, 1, 2, 3, or "not tested". A scoring key of 0 - does not initiate, 1 - initiates, 2 - partially completes, and 3 - completed, is used. Scoring the GMFM-66 requires the use of a computer program called the Gross Motor Ability Estimator (GMAE). Individual item scores are entered and a mathematical algorithm calculates an interval level total score. The total score is an estimate of the child's gross motor function. The range of total score in GMFM-66 is from 0 to 100. The range of % in GMFM-88 is from 0 to 100. Higher values represent a better outcome.
Time Frame: Change in baseline Gross Motor Function Measure 66 at 16weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
scores on a scale | 2.24 (2.32) | 0.81 (0.97)

6. Secondary Outcome: Change of Physical Activity(Steps)
Description: Steps(counts) was measured during the day using ActiGraph(model GT3X, ActiGraph, Pensacola, FL, USA)
Time Frame: Change in baseline steps at 16weeks
Measure: Mean (Standard Deviation); unit: step counts per minute
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
step counts per minute | -37.97 (140.50) | 20.94 (180.53)

7. Secondary Outcome: Change of Resting Heart Rate(RHR)
Description: Resting heart rate(beats/min) is a category of physical fitness, which is measured during graded submaximal exercise test. A normal resting heart rate for adults ranges from 60 to 100 beats per minute. Generally, a lower heart rate at rest implies more efficient heart function and better cardiovascular fitness.
Time Frame: Change in baseline resting heart rate at 16weeks
Population: Participants want to stop during measurement (Intervention group -> 3 participants; Control group -> 2 participants)
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 21
beats per minute | -12.40 (11.98) | -0.62 (8.41)

8. Secondary Outcome: Change of Respiratory Exchange Ratio(RER)
Description: All patients performed a symptom-limited, treadmill exercise test using the Modified Naughton protocol. Respiratory exchange ratio(RER) were measured with a gas analyzer. RER is the ratio between the amount of carbon dioxide (CO2) produced in metabolism and oxygen (O2) used. A high RER (RER values≥1) indicates that carbohydrates are being predominantly used, whereas a low RER (RER values<1) suggests lipid oxidation.
Time Frame: Change in baseline respiratory exchange ratio at 16weeks
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 21
Ratio | 0.04 (0.05) | 0.01 (0.05)

9. Secondary Outcome: Change of Heart Rate Recovery(HRR)
Description: All patients performed a symptom-limited, treadmill exercise test using the Modified Naughton protocol. In the recovery period, the patients walked for 2 minutes at a speed of 1.9 km/h and a grade of 0% and then sat down in a chair for the last 3 minutes (recovery). The Heart rate recovery (HRR) was defined as the difference between peak HR during the test and HR at 1 (HRR1), 3 (HRR3), and 5 (HRR5) minutes.
Time Frame: Change in baseline heart rate recovery at 16weeks
Measure: Mean (Standard Deviation); unit: beats per minute
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 13 | 13
beats per minute
  Change of heart rate recovery 1 | 6.54 (6.34) | -2.15 (5.20)
  Change of heart rate recovery3 | 13.38 (12.92) | -5.54 (5.81)
  Change of heart rate recovery5 | 11.15 (11.42) | -3.80 (7.07)

10. Secondary Outcome: Change of Children Health Questionnaire Parent Form 50 (CHQ-PF50)
Description: The Child Health Questionnaire™ (CHQ) is a family of generic person-reported outcomes measures to assess health-related quality of life for children and adolescents from 5-to-18 years of age. Child Health Questionnaire Parent Form 50 (CHQ-PF50) Questions; total 50 questions, 4 or 6 score Likert scale, the score range is from 0 to 100, higher values represent a better outcome. Scores can be analyzed at combined to derive an overall physical and psychosocial score, (CHQ Summary Scores).
Time Frame: Change in baseline child health questionnaire-parent form 50 at 16weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
score on a scale
  Summary score(Physical) | 2.73 (7.42) | 2.08 (7.78)
  Summary score(Psychosocial) | 3.31 (7.78) | 2.50 (6.65)

11. Secondary Outcome: Change of Timed up and go(TUG)
Description: ① Stand up from the chair without support. ② Walk 3m from chair. ③ Turn around. ④ Sit back in the chair. Measure the time(second), higher values represent a worse outcome. Lower values represent a better outcome.
Time Frame: Change in baseline timed up and go at 16weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
seconds | -1.55 (1.19) | -1.33 (3.64)

12. Secondary Outcome: Change of 6 Minute Walk Test(6MWT)
Description: The 6 minute walk test assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity and endurance. Higher values represent a better outcome.
Time Frame: Change in baseline 6 minute walk test at 16weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
meters | 37.22 (49.52) | 13.43 (37.47)

13. Secondary Outcome: Change of Blood Pressure(BP)
Description: Blood pressure(mmHg) measured before graded exercise test using treadmill.
Time Frame: Change in baseline blood pressure at 16weeks
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 20 | 21
mmHg
  Change of SBP | -1.30 (7.03) | 0.05 (6.29)
  Change of DBP | -1.55 (8.22) | 0.52 (7.73)

14. Secondary Outcome: Change of Pediatric Balance Scale(PBS)
Description: PBS is a functional balance scale adapted and customized from Berg Balance Scale for use with children. The PBS has been used initially to measure the balance functions for school-age children with mild-to-moderate motor impairments. The PBS is a 14-item, criterion-referenced measure, which examines functional balance in the context of everyday tasks. It can easily be administered and scored in less than 20 minutes using equipment commonly found in schools and clinics. Scoring (0-4) is based on how long a specific movement or position is performed, how long the position can be maintained, or how much assistance it requires. The range of total score is from 0 to 56. Higher values represent a better outcome.
Time Frame: Change in baseline pediatric balance scale at 16weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
score on a scale | 2.48 (2.00) | 0.30 (0.88)

15. Secondary Outcome: Change of Attention Deficit Hyperactivity Disorder (ADHD) Rating Scale
Description: ADHD(attention deficit hyperactivity disorder) rating scale; total 18 questions. Each item is scored from 0-3 points, The treatment effect is evaluated using Total score(0 ~ 54 points),attention-deficit scores (0 ~ 27 points) and hyperactivity/impulsivity score (0 ~ 27 points)
Time Frame: Change in baseline ADHD rating scale at 16weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
score on a scale
  Total score(pre) | 12.22 (8.66) | 11.13 (8.32)
  Total score(post) | 11.17 (8.32) | 10.26 (8.20)

16. Secondary Outcome: Change of Self-Esteem Scale
Description: Self-Esteem Scale; total 10 question, Each item is scored from 1-4 points. Five of the ten questions are positive and five are negative. In the positive item, 1 = 'almost not so' and 4 = 'always'. In the negative item, the scores range from 10 to 40. The treatment effect is evaluated using the total score.
Time Frame: Change in baseline self-esteem at 16weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
score on a scale
  Pre-test outcome | 31.22 (4.34) | 32.48 (2.81)
  Post-test outcome | 32.35 (3.61) | 33.34 (3.72)

17. Secondary Outcome: Change of PedsQL 4.0
Description: PedsQL 4.0; total 23 questions; Each item is scored from 0-4 points and scores are transformed on a scale from 0 to 100. Items are reversed scored and linearly transformed to a 0-100 scale as follows: 0=100, 1=75, 2=50, 3=25, 4=0. Thus, the scores range from 0 to 2300, higher values represent a better outcome.
Time Frame: Change in baseline quality life of child at 16weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
score on a scale
  Physical functioning(pre) | 60.73 (19.21) | 65.90 (18.15)
  Physical functioning(post) | 69.70 (15.81) | 77.85 (15.10)
  Emotional functioning(pre) | 70.22 (24.84) | 69.57 (27.67)
  Emotional functioning(post) | 79.13 (20.49) | 82.17 (16.98)
  Social functioning(pre) | 58.48 (28.14) | 61.30 (27019)
  Social functioning(post) | 74.13 (16.90) | 80.65 (22.02)
  School functioning(pre) | 69.35 (22.98) | 72.39 (24.67)
  School functioning(post) | 74.13 (18.99) | 85.44 (12.33)

18. Secondary Outcome: Change of Continuous Performance Test 3rd Edition
Description: Continuous Performance Test 3rd edition; It is a computerized assessment tool designed to measure attention-related problems, instructing them to respond to all stimuli except alphabet X, and instructing them to perform as accurately and quickly as possible. Detectability, Omission Errors, Commission Errors, Perseverations, HRT(hit reaction time), HRT SD (standard deviation), Variability, HRT Block Change, HRT ISI Change are used to assess respondents' performance on inattentiveness, impulsivity, sustained attention, and vigilance. It is used 9 T-scores to assess the level of attention problem.
Time Frame: Change in baseline attention at 16weeks
Measure: Mean (Standard Deviation); unit: T-scores
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
T-scores
  detectability(pre) | 59.00 (7.62) | 54.00 (7.76)
  detectability(post) | 52.57 (10.23) | 49.61 (8.11)
  Omissions(pre) | 71.70 (16.66) | 59.91 (11.29)
  Omissions(post) | 67.13 (18.61) | 57.91 (14.84)
  Commisions(pre) | 48.74 (9.90) | 46.65 (9.47)
  Commisions(post) | 42.96 (7.50) | 43.13 (7.24)
  Perseveration(pre) | 61.30 (13.65) | 51.57 (8.77)
  Perseveration(post) | 53.04 (8.22) | 49.91 (6.82)
  hit reaction time(pre) | 69.87 (14.75) | 65.04 (11.31)
  hit reaction time(post) | 70.04 (14.22) | 65.70 (12.31)
  standard deviation of hit reaction time(pre) | 65.74 (12.08) | 55.83 (10.18)
  standard deviation of hit reaction time(post) | 60.78 (12.14) | 55.04 (9.77)

19. Secondary Outcome: Change of Quantitative Electroencephalography
Description: An electroencephalogram (EEG) is a test that detects electrical activity in your brain using small, metal discs(electrodes) attached to your scalp. Your brain cells communicate via electrical impulses and are active all the time. This activity shows up as wave lines on an EEG recording. It is using Neuroscan Synamp2 amplifier(Compumedics USA, El Paso, TX, USA). For quantitative analysis, EEG without a handwriting is digitized by Fast Fourier Transformation. The square root of the magnitude of the EEG was calculated as the microvolt (uV) value, and the relative power is defined as the electrical force of the specific region divided by the electrical force in the whole region. The relative power of delta, theta, alpha, and beta waves and theta/beta ratio measured at the Fz, Cz, Pz electrode are used for the analysis. The value of theta/beta ratio is average as it approaches 0 and deviates from the mean as it gets away from 0.
Time Frame: Change in baseline Quantitative electroencephalography at 16weeks
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Intervention Group | Control Group
Number analyzed (Participants) | 23 | 23
Z-score
  Fz(pre) | 0.384 (0.961) | -0.046 (0.910)
  Fz(post) | 0.522 (0.835) | -0.098 (0.826)
  Cz(pre) | 0.501 (1.420) | 0.058 (0.883)
  Cz(post) | 0.274 (0.933) | 0.342 (0.760)
  Pz(pre) | 0.077 (0.857) | -0.130 (0.980)
  Pz(post) | 0.240 (1.141) | -0.156 (0.730)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Hippotherapy were conducted by three therapeutic riding instructors. One leader and two side walkers walked with a horse, and all participants wore helmets. The intensity of the exercises and degree of assistance were individualized according to the participants' ability to control their body and horse. The horse/ponies were very experienced in Hippotherapy settings.
Arm/Group | Intervention Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-26): https://cdn.clinicaltrials.gov/large-docs/93/NCT03870893/Prot_SAP_000.pdf